CLINICAL TRIAL: NCT00493246
Title: A Prospective, Multi-Center, Randomized, Open-Label, Single and Repeated Dose, 48 Hour Study, of Intravenous Acetaminophen in Pediatric Inpatients to Determine Pharmacokinetics (PK) and Safety in Acute Pain and Fever
Brief Title: Safety and Pharmacokinetic (PK) Study of Intravenous (IV) Acetaminophen Administration in Pediatric Inpatients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPI-APA-102
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Results first posted 2010-12-29 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Pain; Fever
MeSH Terms: conditions — Pain; Fever | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous (IV) Acetaminophen 15 milligrams/kilogram (mg/kg) (Experimental): Intravenous Acetaminophen administered 15 milligrams/kilogram (mg/kg) every 8 hours (q8h) or every 6 hours (q6h) based age of subject
  Interventions: Drug: IV Acetaminophen
- Intravenous (IV) Acetaminophen 12.5 (mg/kg) (Experimental): Intravenous Acetaminophen administered 12.5 milligrams/kilogram (mg/kg) every 6 hours (q6h) or every 4 hours (q4h)
  Interventions: Drug: IV Acetaminophen

INTERVENTIONS:
Drug: IV Acetaminophen — This study will investigate two doses (12.5 milligrams/kilogram (mg/kg) and 15 milligrams/kilogram) based on weight administered every four hours (q4h), every six hours (q6h), or every eight hours (q8h) (depending on age)
  Neonates: 12.5 mg/kg q6h IV acetaminophen Neonates: 15 mg/kg q8h IV acetaminophen Infants: 12.5 mg/kg q4h IV acetaminophen Infants: 15 mg/kg q6h IV acetaminophen Children: 12.5 mg/kg q4h IV acetaminophen Children: 15 mg/kg q6h IV acetaminophen Adolescents: 12.5 mg/kg q4h IV acetaminophen Adolescents: 15 mg/kg q6h IV acetaminophen
  Other Names: APAP; IV APAP
  Arms: Intravenous (IV) Acetaminophen 12.5 (mg/kg)
Drug: IV Acetaminophen — This study will investigate two doses (12.5 milligrams/kilogram (mg/kg) and 15 milligrams/kilogram) based on weight administered every four hours (q4h), every six hours (q6h), or every eight hours (q8h) (depending on age)
  Neonates: 12.5 mg/kg q6h IV acetaminophen Neonates: 15 mg/kg q8h IV acetaminophen Infants: 12.5 mg/kg q4h IV acetaminophen Infants: 15 mg/kg q6h IV acetaminophen Children: 12.5 mg/kg q4h IV acetaminophen Children: 15 mg/kg q6h IV acetaminophen Adolescents: 12.5 mg/kg q4h IV acetaminophen Adolescents: 15 mg/kg q6h IV acetaminophen
  Other Names: APAP; IV APAP
  Arms: Intravenous (IV) Acetaminophen 15 milligrams/kilogram (mg/kg)

SUMMARY:
We are doing this study to find out what happens to acetaminophen in the body after it is given to children through the vein. Children's bodies may handle drugs differently than adults. Understanding how long the drug stays in the body and how the drug is changed or metabolized by the body (called pharmacokinetics) is an important step in learning what the best dose of acetaminophen for children should be. We are also interested in learning about the safety of this medication when given to children.

DETAILED DESCRIPTION:
A Prospective, Multi-Center, Randomized, Open-Label, Single and Repeated Dose, 48 Hour Study, of Intravenous Acetaminophen in Pediatric Inpatients to Determine Pharmacokinetics (PK) and Safety in Acute Pain and Fever

ELIGIBILITY:
To be eligible for entry into the Study, Subjects must meet or Subjects' Parent or Guardian must meet, agree with or confirm all of the following criteria:

1. Provide written Informed Consent/Assent prior to participation in the Study
2. Age strata:

   * Full-term Neonates (≤ 28 days old and minimum post conception age of 37 weeks at birth)
   * Infants [29 days to <2 years (yrs) old]

     * 29 days to <6 months
     * 6 to <12 months
     * 12 to <24 months)
   * Children (2 yrs to <12 yrs old)
   * Adolescents (12 yrs to ≤16 yrs old)
3. Inpatient status: are currently inpatients or have an admission scheduled and will soon become an inpatient (e.g., elective surgery)
4. Diagnosis: requires or will require analgesic treatment for acute pain or antipyretic treatment for fever
5. IV access: have a need for IV access for the duration of the Study either due to a nothing by mouth (NPO) status or due to the Investigator's assessment that oral treatment is not optimal (for example, severe nausea or vomiting)
6. The Subject's Parent/Guardian must have the ability to read and understand the Study procedures and have the ability to communicate meaningfully with the Study Investigator and staff
7. Be free of other physical, mental, or medical conditions which, in the opinion of the Investigator after completing the screening assessment, make Study participation inadvisable
8. If a female of child bearing potential, have a negative pregnancy test

Exclusion Criteria (Screening)

A Subject is NOT eligible for entry if ANY of the following criteria are met:

1. Is not able to comply with the plasma sampling requirements of the Study
2. Has known or suspected hypersensitivity to acetaminophen or the inactive excipients of IV Acetaminophen.
3. Has been taking any acetaminophen-containing product in the 12 hours prior or any of the following in the 48 hours prior to randomization in the Study: probenecid, disulfiram, isoniazide, St. John's wort, skullcap, chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, and valerian
4. Has any significant medical condition that in the opinion of the Investigator contraindicates participation in the Study
5. Has impaired liver function, with evidence of clinically significant liver disease, or other condition that may suggest the potential for an increased susceptibility to hepatic toxicity with IV APAP exposure. For this criterion, a total bilirubin greater than 1.5 times upper limit of normal (ULN) for age or an Alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) or Aspartate transaminase (AST) serum glutamic oxaloacetic transaminase (SGOT) greater than 2.5 times ULN for age will be deemed as evidence of clinically significant (Common Terminology Criteria for Adverse Events [CTCAE] Grade 2) liver dysfunction or disease.
6. Has significantly impaired renal function or known significant renal disease, as evidenced by an estimated glomerular filtration rate (using the Schwartz formula) calculated to be less than 1/3rd of normal for the applicable age strata
7. Has participated in another interventional clinical Study (investigational or marketed product) within 30 days of the planned Study randomization date

Ages: 29 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Lucile Packard Children's Hospital, Stanford, California
  - CS Mott Childrens Hospital, Ann Arbor, Michigan
  - Duke University Health Systems, Durham, North Carolina
  - Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital Of Pittsburgh, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 sites in the US from 27 June 2007 to 01Sep 2008.
Groups:
- Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen: Full term neonates, 12.5 milligram(mg)per kilogram (kg) IV acetaminophen administered every 6 hours (q6h) (max daily dose of 50 mg/kg)
- Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen: Full term neonates, 15 milligrams (mg)/kilogram (kg) Intravenous(IV) acetaminophen administered every 8 hours (q8h) (max daily dose of 50 mg/kg)
- Infants: 12.5 mg/kg q4h IV Acetaminophen: Infants aged 29days to less than 24months received IV acetaminophen 12.5 mg/kg every 4 hours (q4h)(maximum of 660 mg/dose). Total maximum daily dose is 75 mg/kg or 4 grams, whichever is less.
- Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen: Infants aged 29days to less than 24months received IV acetaminophen 15 mg/kg every 6 hours (maximum dose of 1 gram) Total maximum daily dose is 75 mg/kg or 4 grams, whichever is less.
- Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen: Children aged 2 years to less than 12 years received IV acetaminophen 12.5 mg/kg every 4 hours(maximum of 660 mg/dose). Total maximum daily dose is 75 mg/kg or 4 grams, whichever is less.
- Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen: Children aged 2 years to less than 12 years received IV acetaminophen 15 mg/kg every 6 hours (maximum dose of 1 gram) Total maximum daily dose is 75 mg/kg or 4 grams, whichever is less.
- Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen; Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen: Adolescents aged 12 years to less than or equal to 16 years received IV acetaminophen 15 mg/kg every 6 hours (maximum dose of 1 gram) Total maximum daily dose is 75 mg/kg or 4 grams, whichever is less.
Period: Overall Study
Arm/Group | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen | Infants: 12.5 mg/kg q4h IV Acetaminophen | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen
Started | 2 | 1 | 12 | 13 | 9 (All subjects who were randomized.Excludes 1 subject who was randomized in error.) | 16 (All subjects who were randomized.) | 12 (All subjects who were randomized.) | 10 (All subjects who were randomized.)
Completed | 2 (Completed study 30 days after the last dose) | 1 (Completed study 30 days after the last dose) | 12 (Completed study 30 days after the last dose) | 13 (Completed study 30 days after the last dose) | 8 (Completed study 30 days after the last dose) | 15 (Completed study 30 days after the last dose) | 11 (Completed study 30 days after the last dose) | 10 (Completed study 30 days after the last dose)
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — No access to draw blood | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen | Infants: 12.5 mg/kg q4h IV Acetaminophen | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Total
Number analyzed (Participants) | 2 | 1 | 12 | 13 | 9 | 16 | 12 | 10 | 75
Age, Categorical [Count of Participants; unit: Participants] — The Safety Population (subjects who received any part of a dose of IV acetaminophen) are included in this baseline measure.
  Participants
    <=18 years | 2 | 1 | 12 | 13 | 9 | 16 | 12 | 10 | 75
    Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — The Safety Population (subjects who received any part of a dose of IV acetaminophen) are included in this baseline measure.
  Participants
    Female | 1 | 1 | 4 | 7 | 4 | 6 | 2 | 6 | 31
    Male | 1 | 0 | 8 | 6 | 5 | 10 | 10 | 4 | 44

OUTCOME MEASURES:

1. Primary Outcome: Single-dose Maximum Plasma Concentration (Cmax) , Micrograms Per Milliliter (µg/mL) Pharmacokinetics of IV Acetaminophen
Description: Cmax: Maximum Plasma Concentration
Time Frame: Time Zero (just prior to first dose) to 24 hours post first dose
Population: Subjects who received at least one dose of IV acetaminophen and had at least 3 PK sampling assessments were included in the PK analysis.This outcome measure represents PK parameters for the first dose of IV acetaminophen.
Measure: Median (Full Range); unit: micrograms per milliliter (µg/mL)
Arm/Group | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen | Infants: 12.5 mg/kg q4h IV Acetaminophen | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen
Number analyzed (Participants) | 2 | 1 | 12 | 13 | 9 | 16 | 12 | 10
micrograms per milliliter (µg/mL) | 40.1 [15.9 to 64.4] | 20.1 [20.1 to 20.1] | 16.7 [12.1 to 23.0] | 19.3 [16.2 to 25.4] | 18.2 [13.5 to 27.1] | 21.6 [14.4 to 60.8] | 15.9 [10.6 to 28.8] | 25.5 [9.91 to 49.8]

2. Primary Outcome: Single-dose Time to Reach Maximum Plasma Concentration [Tmax(h)] Pharmacokinetics of IV Acetaminophen
Description: Tmax: Time to reach maximum plasma concentration (Cmax)
Time Frame: Time Zero (just prior to first dose) to 24 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen | Infants: 12.5 mg/kg q4h IV Acetaminophen | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen
Number analyzed (Participants) | 2 | 1 | 12 | 13 | 9 | 16 | 12 | 10
Hour | 0.450 [0.400 to 0.500] | 0.333 [0.333 to 0.333] | 0.267 [0.000 to 0.383] | 0.267 [0.250 to 0.933] | 0.250 [0.0833 to 0.300] | 0.250 [0.0833 to 0.417] | 0.250 [0.0833 to 0.283] | 0.267 [0.00 to 0.333]

3. Primary Outcome: Multiple-dose Area Und the Curve (AUC) From Time 0 (Predose) to the Time of the Dosing Interval at Steady-state (0-t (µg*h/ml) Pharmacokinetics of IV Acetaminophen
Description: AUC 0-t (µg*h/ml): Area under the plasma concentration versus time curve from time 0 (predose) to the time of the dosing interval at steady-state.
Time Frame: Time Zero (just prior to first dose) to 48 hours post first dose
Measure: Median (Full Range); unit: µg*h/ml
Arm/Group | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen | Infants: 12.5 mg/kg q4h IV Acetaminophen | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen
Number analyzed (Participants) | 2 | 1 | 12 | 13 | 9 | 16 | 12 | 10
µg*h/ml | 65.6 [55.8 to 75.4] | 105 [105 to 105] | 43.3 [9.15 to 79.2] | 51.9 [36.0 to 200] | 37.8 [11.3 to 52.3] | 48.0 [32.2 to 131] | 47.7 [22.4 to 132] | 64.0 [33.2 to 84.1]

4. Primary Outcome: Multiple-dose Terminal Elimination Half-life [t1/2(h)] Pharmacokinetics of IV Acetaminophen
Description: t1/2: Terminal elimination half-life
Time Frame: 48hrs
Population: Subjects who received at least one dose of IV acetaminophen and had at least 3 PK sampling assessments were included in the PK analysis.This outcome measure represents PK parameters for the last dose of IV acetaminophen.
  Due to only one subject in the Neonate 15mg/kg group, t1/2 (h) was not calculated.
Measure: Median (Full Range); unit: Hours
Arm/Group | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen | Infants: 12.5 mg/kg q4h IV Acetaminophen | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen
Number analyzed (Participants) | 2 | 0 | 12 | 13 | 9 | 16 | 12 | 10
Hours | 3.88 [3.88 to 3.88] |  | 2.37 [1.15 to 2.81] | 2.79 [2.10 to 5.43] | 2.64 [2.24 to 4.46] | 2.77 [2.15 to 4.85] | 3.37 [2.69 to 4.16] | 4.10 [2.48 to 4.36]

5. Secondary Outcome: Number of Subjects Reporting at Least One Treatment-Emergent Adverse Event (TEAE)
Description: A TEAE is defined as an adverse event that starts on or after the start of study medication
Time Frame: First dose of study medication to 30 days after the last dose of study medication
Measure: Number; unit: Participants
Arm/Group | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen | Infants: 12.5 mg/kg q4h IV Acetaminophen | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen
Number analyzed (Participants) | 2 | 1 | 12 | 13 | 9 | 16 | 12 | 10
Participants | 2 | 1 | 10 | 9 | 2 | 11 | 10 | 6

6. Secondary Outcome: Subjects Who Experience at Least One Serious Treatment-Emergent Adverse Event (TEAE)
Description: A Serious Treatment Emergent Adverse Event is defined as any untoward medical occurrence at any dose of IV acetaminophen that; Results in Death, Is life-threatening, Requires inpatient hospitalization or causes prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, Is a congenital anomaly/birth defect, Is an important medical event
Time Frame: First dose to 30 days following last dose of study medication
Population: All analyses of safety were conducted on the Safety population, which included those subjects who received any portion of a dose of IV acetaminophen.
Measure: Number; unit: Participants
Arm/Group | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen | Infants: 12.5 mg/kg q4h IV Acetaminophen | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen
Number analyzed (Participants) | 2 | 1 | 12 | 13 | 9 | 16 | 12 | 10
Participants | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were reported from the start of study medication to 30 days following the last dose of study medication.
Arm/Group | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen | Infants: 12.5 mg/kg q4h IV Acetaminophen | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/12 | 1/13 | 1/9 | 2/16 | 1/12 | 1/10
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 10/12 | 7/13 | 1/9 | 10/16 | 10/12 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen (N=2) | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen (N=1) | Infants: 12.5 mg/kg q4h IV Acetaminophen (N=12) | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen (N=13) | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen (N=9) | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen (N=16) | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen (N=12) | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen (N=10)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mediastinal disorders chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural drainage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thoracic cavity drainage test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neonates:12.5 mg/kg Every 6 Hours (q6h) IV Acetaminophen (N=2) | Neonates: 15 mg/kg Every 8 Hours (q8h) IV Acetaminophen (N=1) | Infants: 12.5 mg/kg q4h IV Acetaminophen (N=12) | Infants:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen (N=13) | Children: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen (N=9) | Children: 15 mg/kg Every 6 Hours(q6h) IV Acetaminophen (N=16) | Adolescents: 12.5 mg/kg Every 4 Hours (q4h) IV Acetaminophen (N=12) | Adolescents:15 mg/kg Every 6 Hours (q6h) IV Acetaminophen (N=10)
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 0 | 3 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Central Line Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular Spasm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0
Face edema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 0 | 1 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 5 | 2
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0 | 0 | 3 | 1 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural Hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 5 | 1 | 2
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Vocal Cord Paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Median ranges were not calculated or not assessable for neonates at the following due to limited samples.:

* 12.5 mg/kg q6h- t1/2 (h)
* 15 mg/kg q8h -Cmax, Tmax, AUC0-t and t1/2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may publish 18 months after Cadence's final evaluation of all study data from all sites, whichever occurs first.Manuscripts/abstracts will be provided to Cadence for review and comment at least 30 days prior to submission.Cadence shall have 30 days to respond with comments.